CLINICAL TRIAL: NCT04030546
Title: Ivabradine to Prevent Anthracycline-induced Cardiotoxicity: a Prospective Randomized Open Label Clinical Trial
Brief Title: Ivabradine to Prevent Anthracycline-induced Cardiotoxicity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Sigita Aidietiene, Assoc. Prof., Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICO
Record Dates: First submitted 2019-07-22; First posted 2019-07-24 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-07

CONDITIONS: Patients With Cancer
Keywords: anthracycline chemotherapy; cardiotoxicity; heart failure
MeSH Terms: conditions — Cardiotoxicity; Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ivabradine (Active Comparator): Patients will receive ivabradine just before anthracycline chemotherapy, 5 mg per oral twice daily, until the last chemotherapy session
  Interventions: Drug: Ivabradine
- Usual care (No Intervention): Patient will receive usual care

INTERVENTIONS:
Drug: Ivabradine — Ivabradine capsule
  Arms: Ivabradine

SUMMARY:
The aim of this study is to investigate protective effects of ivabradine in adult cancer patients undergoing anthracycline-based chemotherapy.

DETAILED DESCRIPTION:
Cancer treatment with anthracyclines may cause heart damage and can lead to heart failure. There are drugs which may protect against cardiotoxic effects of anthracyclines (renin-angiotensin inhibitors and beta blockers), but they are not tolerated due to hypotension. Ivabradine is heart rate lowering drug without effect on blood pressure which was approved for treatment of angina pectoris and heart failure. The aim of this study is to investigate protective effects of ivabradine in cancer patients undergoing anthracycline-based chemotherapy.

Ivabradine selectively inhibits If currents in the sinus node and prolongs the duration of spontaneous depolarization. That controls the heart's contractions and regulates the heart rate. Additionally, ivabradine might preserve myocardial function and contractility without effect on blood pressure. Ivabradine was approved for symptomatic treatment of chronic stable angina pectoris and chronic heart failure.

The aim of this study is to investigate protective effects of ivabradine in adult cancer patients undergoing anthracycline-based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients undergoing anthracyclines based chemotherapy;
* heart rate (HR) > 70 times per minute;
* Written informed consent.

Exclusion Criteria:

* Contraindications for ivabradine administration;
* HR<70 times per minute;
* Incapability to complete informed consent;
* Severe valve disease;
* Left ventricular ejection fraction (LVEF)≤ 30 %;
* Other severe conditions;
* Poor echogenicity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in left venticular dysfunction by global longitudinal strain (GLS). | 1, 3 and 6 months
  Change in global longitudinal strain (GLS) at least by 3%.

SECONDARY OUTCOMES:
Incidence of myocardial injury according to levels of high-sensitivity cardiac troponin T and NT-proBNP | 1, 3 and 6 months
  Incidence of myocardial injury according to levels of high-sensitivity cardiac troponin T and NT-proBNP.
Incidence of left ventricular systolic and diastolic dysfunction by 2D and 3D echocardiography. | 1, 3 and 6 months
  Incidence of left ventricular (LV) dysfunction defined as drop of LV ejection fraction by ≥ 10%.

OTHER OUTCOMES:
Incidence of symptomatic heart failure. | 1, 3 and 6 months
  Incidence of symptomatic heart failure.
Changes in left ventricular and right ventricular dimensions by 2D and 3D echocardiography. | 1, 3 and 6 months
  Changes in left ventricular and right ventricular dimensions by 2D and 3D echocardiography.

CONTACTS AND LOCATIONS:
Overall Officials: Sigita Aidietiene, MD, PhD, Principal Investigator — Vilnius University
Locations (1):
- Vilnius University Hospital Santaros klinikos, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No